CLINICAL TRIAL: NCT06767592
Title: A Single-Arm Open-Label Feasibility Study of Probiotics for the Modulation of the Gut Microbiome in IgA Nephropathy (Pro-IgAN)
Brief Title: A Study of Probiotics in IgA Nephropathy
Acronym: Pro-IgAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: Kidney Cancer UK (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0718
Record Dates: First submitted 2023-10-09; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Probiotic (Experimental): Participants will receive the multi-strain probiotic, Bio-Kult Advanced, 2 capsules twice daily between baseline and month 3 visits.
  Interventions: Dietary Supplement: Bio-Kult Advanced

INTERVENTIONS:
Dietary Supplement: Bio-Kult Advanced — Bio-Kult Advanced will be provided as capsules and can be stored at room temperature. Participants will be instructed to swallow two capsules in the morning and two capsules in the evening, with food.

SUMMARY:
IgA nephropathy (IgAN) occurs when a specific form of the IgA antibody lodges on the kidneys and causes damage, which may lead to kidney failure. This form of IgA is likely to come from the gut and the upper airways.

Recent studies have shown that the bacteria that live in these areas may be different in IgAN. We think that the interaction between these and the immune system triggers production of the IgA that leads to kidney damage. We will examine these bacteria in detail, and test whether a probiotic can alter this favorably, and reduce harmful forms of IgA production in IgAN.

DETAILED DESCRIPTION:
The purpose of this proposal is to conduct a proof of concept study, to test the hypothesis that dysbiosis of the gut microbiota plays a critical role in the development of IgAN.

Objectives are firstly, to characterise the gut microbiome, and faecal, plasma and urine metabolome, in relation to biomarkers of mucosal immunity and glomerular disease in patients with IgAN. Secondly, Investigators will test whether a multi-strain probiotic (Bio-Kult Advanced) produces a modulatory effect on these indices. The probiotic has been selected with our industry collaborator Protexin, based on previous studies demonstrating reduced faecal microbial diversity in patients with progressive IgAN, compared to those with non-progressive IgAN and healthy subjects.

This study will further our understanding of the interplay between the gut microbiome, metabolome, and mucosal immune system in IgAN. Investigators will generate important pilot data, to inform the design of a longer-term randomised clinical trial of probiotics in IgAN, and to identify potential plasma biomarkers to highlight those at risk of progressive disease, and those who may respond to treatments targeted to the gut.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven IgAN
2. Age 18 years or older
3. Able and willing to give informed consent
4. Sufficient understanding of English to understand the patient information sheet and complete questionnaires
5. No change in medications for 6 weeks up to the Baseline visit
6. Stable diet (e.g. not a change to elimination, reduction, vegan or vegetarian diet) for 30-days prior to the baseline visit and during the study

Exclusion Criteria:

1. Aged <18 years
2. Unable or unwilling to give informed consent
3. eGFR < 45 ml/min/1.73 m2 (measured by CKD-EPI formula)
4. Already taking a regular pre- or pro-biotic supplement or other dietary supplement aimed at modulating the gut microbiota, within the previous 60-days
5. Predicted to change diet during the study
6. Any of the following conditions:

   6.1. Autoimmune disease (e.g. systemic lupus erythematosus) 6.2. Serious gastro-intestinal illness (including Crohn's disease, ulcerative colitis, chronic liver disease, significant gastrointestinal surgery or cancer, pancreatitis, motility disorder) 6.3. Diagnosed infectious illness within the previous 30-days
7. Prescribed any of the following medication within the previous 60-days 7.1. Antibiotics or anti-viral medications 7.2. Steroids or other immunosuppressive agents
8. Any other condition which in the opinion of the investigator could interfere with the study
9. Enrolled in a clinical trial of an investigational medicinal product
10. Allergy to any component of BioKult Advanced (including milk or soy allergy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in levels of IgA1 O-glycosylation at Month 3 compared to baseline. | 3 months
  The primary outcome, change in circulating IgA O-glycans levels between baseline and 3-months, will be analysed.

SECONDARY OUTCOMES:
Urine protein/creatinine ratio (UP/C) over a 6-month period | Up to Month 6
  Change from baseline in proteinuria, measured by urinary protein/creatinine ratio [UPCR], up to Month 6
eGFR over a 6 month period | Up to Month 6
  Rate of change in eGFR over a 6 month period from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Leicester General Hospital, University Hospitals of Leicester NHS Trust, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No